CLINICAL TRIAL: NCT03233113
Title: Response Prevention or Response Permission? A Randomized Controlled Trial of the "Judicious Use of Safety Behaviors" During Exposure Therapy (Institutional Review Board Title: Overcome Your Spider Phobia)
Brief Title: The Effects of Safety Seeking Behaviors During Exposure Therapy for Adults With Spider Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Society for a Science of Clinical Psychology (Unknown); Association for Behavioral and Cognitive Therapies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0700
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Specific Phobia
Keywords: Exposure therapy; Cognitive-behavioral therapy; Anxiety disorders
MeSH Terms: conditions — Phobia, Specific; Anxiety Disorders | interventions — Implosive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The current study follows a two-arm, parallel group RCT study design. Participants are randomized to either the active control arm (Exposure and Response Prevention) or the experimental arm (Exposure with Judicious Safety Behaviors). Participants are not offered the opportunity to choose their study condition, nor are they provided with an explanation of the difference between their assigned treatment arm and the alternative treatment arm. Randomization was achieved prior to initial participant recruitment via a random number generator with the condition that an equal number of participants be randomized to each condition.
Who Masked: Outcomes Assessor
Masking Description: Pre-determined condition allocation was listed in an Excel spreadsheet and concealed with black cell masking color. Interested individuals who met initial eligibility criteria during a pre-enrollment phone screening were entered in the order of screening in the assignment Excel spreadsheet (that was already masked to conceal condition assignment). Only the participant's therapist viewed the allocated condition immediately prior to the first treatment session by temporarily lifting the cell mask.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure and response prevention (Active Comparator): Exposure therapy with response prevention involves four hour-long individual sessions with a trained exposure therapist. Session 1 involves functional assessment, psychoeducation, presentation of the treatment rationale, and treatment planning. Sessions 2-4 involve a review of the model/treatment rationale, condition-specific reminders about how to prevent engaging in any safety behaviors during exposure, a 30-minute in-vivo exposure trial involving a live tarantula, and post-exposure processing. Session 4 also involves a discussion of relapse prevention strategies.
  Interventions: Behavioral: Exposure therapy
- Exposure with judicious safety behaviors (Experimental): Exposure therapy with judiciously used safety behaviors for spider phobia involves four hour-long individual sessions with a trained exposure therapist. Session 1 involves functional assessment, psychoeducation, presentation of the treatment rationale, and treatment planning. Sessions 2-4 involve a review of the model/treatment rationale, condition-specific reminders about how to strategically incorporate safety behaviors during exposure, a 30-minute in-vivo exposure trial involving a live tarantula, and post-exposure processing. Session 4 also involves a discussion of relapse prevention strategies.
  Interventions: Behavioral: Exposure therapy

INTERVENTIONS:
Behavioral: Exposure therapy — Exposure therapy (i.e., exposure-based cognitive behavioral therapy) for spider phobia according to condition-specific, scripted treatment manuals inspired by evidence-based exposure programs for anxiety/phobias (for both arms: Abramowitz, Deacon, & Whiteside, 20011; Antony, Craske, & Barlow, 1995) as well as the seminal account of the "judicious use of safety behaviors" thesis (for the experimental arm only: Rachman, Radomsky, & Shafran, 2008). Exposure and response prevention involves confronting a live spider while resisting safety-seeking behaviors; exposure with judicious safety behaviors involves strategically using safety behaviors while confronting a live spider.
  Other Names: Cognitive-behavioral therapy for anxiety disorders

SUMMARY:
Exposure-based cognitive-behavioral therapy (i.e., "exposure therapy"), which entails repeated and prolonged confrontation with feared situations/stimuli, is the most effective treatment for anxiety disorders (e.g., arachnophobia). Safety behaviors are actions performed to prevent, minimize, or escape a feared catastrophe and/or associated distress (e.g., wearing thick shoes or gloves when around areas where there might be spiders). It is understood that safety behaviors contribute to the development and maintenance of anxiety disorders; accordingly, patients' safety behaviors are traditionally eliminated as soon as possible during exposure therapy (i.e., "response prevention"). Unfortunately, not everyone who receives exposure therapy benefits from this approach. To address the limitations of exposure's effectiveness, some experts have questioned the clinical convention of response prevention during exposure therapy. Specifically, they propose the "judicious use of safety behaviors": the careful and strategic incorporation of safety behaviors during exposure therapy. The controversial role of permitting safety behaviors during exposure has garnered substantial research attention, yet study findings are mixed. The current study, therefore, was designed to improve upon the methodological limitations of previous related research and examine the relative efficacy of traditional exposure with response prevention (E/RP) and the experimental exposure with the judicious use of safety behaviors (E/JU) in a sample of adults with arachnophobia. In light of previous related research, several hypotheses were made regarding the short- (posttreatment) and long-term (1-month follow-up) treatment effects:

1. Primary outcomes: E/RP participants will demonstrate greater improvement in spider phobia than the E/JU participants along behavioral and self-report symptom measures at follow-up.
2. Secondary outcomes: Treatment acceptability and tolerability will be higher for E/JU participants, relative to E/RP participants, before beginning exposures and at posttreatment, but not at follow-up. In addition, hypothesize that E/RP participants will report greater reductions in peak distress and greater improvements in distress tolerance relative to E/JU participants at follow-up.
3. Additional outcome: Exploratory analyses will be conducted to compare the relative rate of behavioral approach and exposure goal completion between treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Presence of clinically significant spider phobia
* English fluency
* Willingness to attend and audiotape all study sessions

Exclusion Criteria:

* Spider or bee allergies
* Previous trial of exposure-based cognitive-behavioral therapy for any anxiety problem
* Current alcohol or substance use disorder
* Lifetime symptoms of mania or psychosis
* Voluntarily report current suicidal ideation
* Complete 10 or more steps on the behavioral approach task administered at the pre-treatment assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fear of Spiders Questionnaire Score at 1-month follow-up | Baseline, 1-month follow-up
  The Fear of Spiders Questionnaire (FSQ; Szymanski & O'Donahue, 1995) is an 18-item self-report measure of spider phobia. Participants rate their agreement with each statement (e.g., "If I saw a spider now, I would think it will harm me") on a scale of 0 (totally disagree) to 7 (totally agree). Possible total scores range from 0 to 126, such that higher scores indicate greater spider fear.
Change from baseline Spider Behavioral Approach Task Score at 1-month follow-up | Baseline, 1-month follow-up
  The Spider Behavioral Approach Task (BAT) includes 13 rank-ordered steps ranging from standing at the opposite end of a room containing a tarantula enclosed in a closed terrarium covered with a sheet to allowing the tarantula to crawl up one's bare arm. A participant must perform a BAT step for 10 consecutive seconds for the step to count as completed. BAT scores are recorded as the number of the highest step completed.

SECONDARY OUTCOMES:
Change from baseline FSQ Score at 0-48 hours post-treatment | Baseline, Within approximately 48 hours post final treatment
  The FSQ is an 18-item self-report measure of spider phobia that is included in the baseline and post-treatment assessments. The post-treatment assessment is administered immediately post-treatment (at the end of the fourth/final treatment session), although participants with scheduling conflicts may complete the post-treatment assessment during another visit as long as it occurs within 48 hours of the final treatment (4th overall) visit.
Change from baseline Spider BAT Score at 0-48 hours post-treatment | Baseline, Within approximately 48 hours post final treatment
  The Spider BAT, a behavioral measure of spider phobia, is included in the baseline and post-treatment (within 48 hours of the fourth/final treatment session) assessments.
Treatment Acceptability and Adherence Scale Score at Baseline | Baseline
  The Treatment Acceptability and Adherence Scale (TAAS) is a 10-item self-report measure of treatment acceptability and predicted adherence. Participants rate each statement (e.g., "If I participated in this treatment, I would be able to adhere to its requirements") on a 1 (disagree strongly) to 7 (agree strongly) scale. Possible total scores range from 10 to 70, with higher scores indicating greater treatment acceptability/anticipated adherence.
TAAS Score at 0-48 hours post-treatment | Within approximately 48 hours post final treatment
  The TAAS is a 10-item self-report measure of treatment acceptability and predicted adherence. Participants rate each statement (e.g., "If I participated in this treatment, I would be able to adhere to its requirements") on a 1 (disagree strongly) to 7 (agree strongly) scale. Possible total scores range from 10 to 70, with higher scores indicating greater treatment acceptability/anticipated adherence.
TAAS Score at 1-month follow-up | 1-month follow-up
  The TAAS is a 10-item self-report measure of treatment acceptability and predicted adherence. Participants rate each statement (e.g., "If I participated in this treatment, I would be able to adhere to its requirements") on a 1 (disagree strongly) to 7 (agree strongly) scale. Possible total scores range from 10 to 70, with higher scores indicating greater treatment acceptability/anticipated adherence.
Change from baseline BAT Peak Distress Score at 0-48 hours post-treatment | Baseline, Within approximately 48 hours post final treatment
  Immediately after completing each step of the BAT (at the baseline and post-treatment assessments), participants are asked to verbally report their (a) anxiety and (b) disgust, using a scale of 0 (not at all) to 10 (maximum). The highest self-reported values are separately recorded as peak BAT anxiety and peak BAT disgust, which are summed together to form a single peak BAT distress value. The post-treatment assessment is administered immediately post-treatment (at the end of the fourth/final treatment session), although participants with scheduling conflicts may complete the post-treatment assessment during another visit as long as it occurs within 48 hours of the final treatment (4th overall) visit.
Change from baseline BAT Peak Distress Score at 1-month follow-up | Baseline, 1-month follow-up
  Immediately after completing each step of the BAT, participants are asked to verbally report their (a) anxiety and (b) disgust, using a scale of 0 (not at all) to 10 (maximum). The highest self-reported values are separately recorded as peak BAT anxiety and peak BAT disgust, which are summed together to form a single peak BAT distress value.
Change from baseline In-Vivo Distress Tolerance Score at 0-48 hours post-treatment | Baseline, Within approximately 48 hours post final treatment
  Immediately after completing the BAT, participants are asked: "Regardless of how intense your distress was, how well did you tolerate your distress? That is, how well were you able to manage whatever emotions and sensations came up during the exercise, even if they were very strong?" Participants verbally report ratings of state distress tolerance using a 0 (not at all able to tolerate my distress) to 10 (completely able to tolerate my distress) scale. The post-treatment assessment is administered immediately post-treatment (at the end of the fourth/final treatment session), although participants with scheduling conflicts may complete the post-treatment assessment during another visit as long as it occurs within 48 hours of the final treatment (4th overall) visit.
Change from baseline In-Vivo Distress Tolerance Score at 1-month follow-up | Baseline, 1-month follow-up
  Immediately after completing the BAT, participants are asked to verbally report their BAT distress tolerance, using a 0 (not at all able to tolerate my distress) to 10 (completely able to tolerate my distress) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Blakey, M.S., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individuals may contact the primary investigator (Shannon M. Blakey) to request access to the Individual Patient Data (IPD) after the termination of the study and publication of the primary outcomes manuscript.

REFERENCES:
- [Background] Blakey SM, Abramowitz JS. The effects of safety behaviors during exposure therapy for anxiety: Critical analysis from an inhibitory learning perspective. Clin Psychol Rev. 2016 Nov;49:1-15. doi: 10.1016/j.cpr.2016.07.002. Epub 2016 Jul 25. PMID 27475477
- [Background] Rachman S, Radomsky AS, Shafran R. Safety behaviour: a reconsideration. Behav Res Ther. 2008 Feb;46(2):163-73. doi: 10.1016/j.brat.2007.11.008. Epub 2007 Nov 28. PMID 18199423
- [Background] Szymanski J, O'Donohue W. Fear of Spiders Questionnaire. J Behav Ther Exp Psychiatry. 1995 Mar;26(1):31-4. doi: 10.1016/0005-7916(94)00072-t. PMID 7642758